CLINICAL TRIAL: NCT02804334
Title: The Role of Molecules in Blood Cells for Diagnosing Bipolar Disorders
Status: Terminated | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: CellPrint Biotechnology (Other)
Responsible Party: Principal Investigator, Keming Gao, Clinical Director, Mood Disorders Program, UH Cleveland Medical Center, University Hospitals Cleveland Medical Center
Other Study IDs: 02-16-34
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Participants with no current or lifetime psychiatric disorders
  Interventions: Procedure: Psychiatric Questionnaires; Procedure: Blood draw
- Untreated Bipolar Disorder: Participants who meet criteria for current bipolar disorder but who are not currently taking any psychotropic medications
  Interventions: Procedure: Psychiatric Questionnaires; Procedure: Blood draw

INTERVENTIONS:
Procedure: Psychiatric Questionnaires
Procedure: Blood draw

SUMMARY:
The goal of this project is to study ~45 molecules in blood cells that may differentiate patients with bipolar disorder from healthy controls.

DETAILED DESCRIPTION:
There is one study visit for this research protocol. Participants may complete this visit on the day that they sign consent. If there is an upcoming blood draw already scheduled for the participant, within the clinical research trial in which they are enrolled, they may decide to wait until then to receive their blood draw. In addition, if a subject has completed the protocol specific monitoring labs within the past 30 days, either for clinical or research purposes, they do not have to be repeated.

After obtaining the informed consent, all potential research participants will be assessed with a systemic clinical interview and a structured interview with the Mini-International Neuropsychiatric Interview (MINI). Psychiatric assessments will be administered to all participants, both healthy controls and participants diagnosed with bipolar disorder (BD). All eligible participants will also complete a Clinical Record Form. The form includes demographics, previous treatment history, the number of previous episodes, family history, and other historical correlates.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers (Group 1)

For inclusion in this study, subjects must meet all of the following criteria:

1. Able to provide informed consent;
2. Male or female, at least 18 years of age;
3. Physically healthy
4. No current and/or lifetime psychiatric disorder assessed with the MINI for Diagnostic and Statistical Manual-5 (DSM-5);
5. Willing to have blood draw.

Exclusion Criteria for Healthy Volunteers (Group 1)

Any of the following is regarded as a criterion for exclusion from the study:

1. Unwilling to comply with study requirements;
2. Unwilling to have blood draw;
3. Patients with chronic medical conditions such as diabetes, cardiovascular disease, immune diseases, infectious diseases and neurological disorders;
4. Tests positive for illegal substances or prescriptions medications for which participants do not have a valid prescription;
5. Currently pregnant.
6. A lifetime history of a psychiatric disorder

Inclusion Criteria for Untreated Bipolar Subjects (Group 2)

For inclusion in this study, subjects must meet all of the following criteria:

1. Able to provide informed consent;
2. Male or female, at least 18 years of age;
3. Meets current DSM-5 criteria for bipolar type I (BPI) or bipolar type II (BP II) disorder as assessed by the MINI.
4. Depression severity should be measured with Montgomery-Asberg Depression Rating Scale (MADRS). A MADRS total score ≥ 20 is required at Screening Visit/Baseline Evaluation.
5. Has experienced impairment as documented by a score consistent with moderate impairment (4 or more on at least one of the three subscales of the Sheehan Disability Scale (SDS), which includes an assessment of work-life, family-life, and social life (no/mild impairment 0-3, moderate impairment 4-6, severe impairment 7-10)
6. Have not taken any psychotropic medications within the past 4 weeks;
7. Willing to have blood draw.

Exclusion Criteria for Untreated Bipolar Subjects (Group 2)

Any of the following is regarded as a criterion for exclusion from the study:

1. Unwilling to comply with study requirements;
2. Unwilling to have blood draw;
3. Patients with chronic medical conditions such as diabetes, cardiovascular disease, immune diseases, infectious diseases, and neurological disorders;
4. Tests positive for illegal substances or prescriptions medications for which participants do not have a valid prescription;
5. Currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll 70 subjects. Thirty-five subjects will have bipolar I or II and are currently not taking any psychotropic medications and 35 subjects will be healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity of ~45 molecules in blood cells of patients with bipolar I or II disorder versus healthy controls | Day 1
Specificity of ~45 molecules in blood cells of patients with bipolar I or II disorder versus healthy controls | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No